CLINICAL TRIAL: NCT04364698
Title: Observational Cohort of COVID-19 Patients at Raymond-Poincare
Acronym: COVID-RPC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 20SBS-COVID-RPC
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The SARS-CoV-2 infection detected in China in December 2019 is responsible for the current COVID-19 pandemic affecting nearly 1.2 million people worldwide to date. Infection with this virus of the coronavirus family is causing a broad clinical spectrum, the main manifestation of which is an influenza-like condition associated with a pattern of severe hypoxemia pneumonia, and in some cases fatal. Little is known about this pathology, so we propose to carry out an observational cohort of patients treated in our hospital for an SARS-CoV-2 infection.

This cohort should make it possible to clinically, biologically and radiologically characterize the SARS-CoV-2 infections. We will also collect the therapeutic strategies implemented, their possible toxicity and the evolution of the patients.

DETAILED DESCRIPTION:
COVID-19 is a virus belonging to the coronavirus family, which includes a large number of viruses that can cause a wide variety of diseases in humans. The SARS-CoV-2 virus that caused the current COVID-19 pandemic, although widely described in the literature, still has many grey areas. The main clinical manifestation is an influenza-like illness associated with respiratory tract infection that can lead to severe hypoxemic pneumonia with fatal outcomes in 2.3% of cases. The clinical spectrum is not yet very well known, as evidenced by the evidence of anosmia, agueusia, or recent skin manifestations, but also strong suspicion of possible neurological damage. Similarly, it is not yet very well established, apart from certain co-morbidities, which patients are likely to develop serious forms requiring admission to intensive care, as shown by the proportion of patients < 60 years of age admitted to intensive care for ARDS.

Moreover, the question of how to manage these patients still raises many questions, particularly about the type of molecules to be introduced and at what point in the history of the disease. Some of these molecules, such as the Lopinavir/Ritonavir combinations and the Hydroxychloroquine/ Azithromycin combination, are not free of complications, particularly cardiac complications requiring close monitoring by ECGs and repeated dosing, the effectiveness of which has not yet been clearly demonstrated.

In order to better understand this infection, we propose to set up a cohort of patients treated for CoV-2 SARS infection on our site.

Study scheme:

Longitudinal cohort study of patients with confirmed or strongly suspected CoV-2 SARS infection.

ELIGIBILITY:
Inclusion criteria:

* Patient ≥ 18 years old
* SARS-CoV-2 infection confirmed by PCR or strongly suspected on compatible radio-clinical grounds during an epidemic period.

Exclusion criteria:

* Not able to express their opposition
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient ≥ 18 years old SARS-CoV-2 infection confirmed by PCR or strongly suspected on compatible radio-clinical grounds during an epidemic period.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
clinical, biological and radiological characteristics | through study completion, an average of 1 month
  Describe the clinical, biological and radiological characteristics of COVID-19 patients hospitalized in our center.

SECONDARY OUTCOMES:
patients' journey description | through study completion, an average of 1 month
  Describe the patients' journey through our structure.
Treatments effects | through study completion, an average of 1 month
  Describe the clinical course of patients treated with the hydroxychloroquine/azithromycin combination in a compassionate context and the side effects observed.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Bessis, MD, Principal Investigator — Infectious diseases department, Raymond Poincaré Hospital, APHP; Aurelien Dinh, MD, Study Director — Infectious diseases department, Raymond Poincaré Hospital, APHP
Locations (1):
- Department of Infectiology, Raymond Poincaré Hospital, APHP, Garches, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epidemiology Working Group for NCIP Epidemic Response, Chinese Center for Disease Control and Prevention. [The epidemiological characteristics of an outbreak of 2019 novel coronavirus diseases (COVID-19) in China]. Zhonghua Liu Xing Bing Xue Za Zhi. 2020 Feb 10;41(2):145-151. doi: 10.3760/cma.j.issn.0254-6450.2020.02.003. Chinese. PMID 32064853
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Rothan HA, Byrareddy SN. The epidemiology and pathogenesis of coronavirus disease (COVID-19) outbreak. J Autoimmun. 2020 May;109:102433. doi: 10.1016/j.jaut.2020.102433. Epub 2020 Feb 26. PMID 32113704
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Cao B, Wang Y, Wen D, Liu W, Wang J, Fan G, Ruan L, Song B, Cai Y, Wei M, Li X, Xia J, Chen N, Xiang J, Yu T, Bai T, Xie X, Zhang L, Li C, Yuan Y, Chen H, Li H, Huang H, Tu S, Gong F, Liu Y, Wei Y, Dong C, Zhou F, Gu X, Xu J, Liu Z, Zhang Y, Li H, Shang L, Wang K, Li K, Zhou X, Dong X, Qu Z, Lu S, Hu X, Ruan S, Luo S, Wu J, Peng L, Cheng F, Pan L, Zou J, Jia C, Wang J, Liu X, Wang S, Wu X, Ge Q, He J, Zhan H, Qiu F, Guo L, Huang C, Jaki T, Hayden FG, Horby PW, Zhang D, Wang C. A Trial of Lopinavir-Ritonavir in Adults Hospitalized with Severe Covid-19. N Engl J Med. 2020 May 7;382(19):1787-1799. doi: 10.1056/NEJMoa2001282. Epub 2020 Mar 18. PMID 32187464
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204